CLINICAL TRIAL: NCT03996811
Title: The Effectiveness of Home-based Walking Program in Improving Physical Functioning, Cardiovascular Health Index, Negative Emotions, and Quality of Life in Patients With Hemodialysis
Brief Title: The Effectiveness of Home-based Walking Program in Improving Quality of Life in Patients With Hemodialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019-06-003A
Record Dates: First submitted 2019-06-23; First posted 2019-06-25 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Hemodialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Experimental): exercise education: A 12-week regimen of home-based walking exercises, include moderate intensity for 40 min, three times a week on non-dialysis days. We explained the participants how to perform the exercises, according to an instruction manual for the exercise regimen. Participants were instructed that the exercises would be effective only if they reached 40%-60% of the target heart rate, as determined by the Karvonen method, and 12-13 on the RPE.
  Interventions: Other: Exercise education
- usual-care group (No Intervention): Hospital routine care

INTERVENTIONS:
Other: Exercise education — weekly telephone consultations concerning exercise. we discussed whether participants' exercise fulfilled the prescribed intensity, duration, or frequency and whether the participants experienced any adverse effects.
  Arms: exercise group

SUMMARY:
This study will investigate the effectiveness of a rehabilitation program in improving physical functioning, cardiovascular health index, negative emotions, and quality of life in patients with hemodialysis in Taiwan.

Hypothesis:

1. The quality of life in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, and 24th month.
2. The negative emotions in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, and 24th month.
3. The cardiovascular health index in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, and 24th month.
4. The Physical Functioning in exercise group is significant improving than usual-care group at 3rd, 6th, 12th, and 24th month.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of a rehabilitation program in improving Physical Functioning, cardiovascular health index, negative emotions, and quality of life in patients with hemodialysis in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

-Patients with hemodialysis who were aged ≥20 years, could communicate in either Mandarin or Taiwanese, 6-minute walking test ≧ 300m and not cognitively impaired were included.

Exclusion Criteria:

-

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-06-24 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
subjective quality of life | 3rd month after recruited
  using Kidney Disease Quality of Life Questionnaire-36™ (KDQOL-36™) to measure quality of life.
subjective quality of life | 6rd month after recruited
  using Kidney Disease Quality of Life Questionnaire-36™ (KDQOL-36™) to measure quality of life.
subjective quality of life | 12rd month after recruited
  using Kidney Disease Quality of Life Questionnaire-36™ (KDQOL-36™) to measure quality of life.
subjective quality of life | 24rd month after recruited
  using Kidney Disease Quality of Life Questionnaire-36™ (KDQOL-36™) to measure quality of life.

SECONDARY OUTCOMES:
subjective negative emotions | 3rd month after recruited
  negative emotions including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
subjective negative emotions | 6rd month after recruited
  negative emotions including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
subjective negative emotions | 12rd month after recruited
  negative emotions including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
subjective negative emotions | 24rd month after recruited
  negative emotions including anxiety and depression (Hospital Anxiety and Depression Scale). The Hospital Anxiety and Depression Scale include anxiety and depression subscales, a total of 7 questions, each subscale is a four-point scoring method, 0 point for "not at all", 3 points for "always do", each subscale scores is between 0 and 21, that a score of 7 or less for non-cases, scores of 8-10 for doubtful cases and scores of 11 or more for definite cases.
objective cardiovascular health index | 3rd month after recruited
  serum
objective cardiovascular health index | 6rd month after recruited
  serum
objective cardiovascular health index | 12rd month after recruited
  serum
objective cardiovascular health index | 24rd month after recruited
  serum
check Physical Functioning | 3rd month after recruited
  6MWT(Six Minute Walk Test)
check Physical Functioning | 6rd month after recruited
  6MWT(Six Minute Walk Test)
check Physical Functioning | 12rd month after recruited
  6MWT(Six Minute Walk Test)
check Physical Functioning | 24rd month after recruited
  6MWT(Six Minute Walk Test)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Mei Chen, PhD, Principal Investigator — National Taipei University of Nursing and Health Sciences; Hsin-Ling Tai, Master, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Jiu-Yun Tian, University, Study Director — Taipei Veterans General Hospital, Taiwan
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (learned intermediary) identified for this purpose.